CLINICAL TRIAL: NCT04501224
Title: The Efficacy and Safety of Tenofovir Alafenamide Fumarate Compared With Other Nucleoside Analogues (Acid) to Treat Patients With Low-level Viremia of HBV
Brief Title: The Efficacy and Safety of TAF vs Other NAs in Patients With LVL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yuehua Huang, Laboratory director of hepatology#Deputy director of infection, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAF
Record Dates: First submitted 2020-07-19; First posted 2020-08-06 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Chronic Hepatitis b; Cirrhosis Due to Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide; entecavir; Tenofovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- switch to tenofovir alafenamide fumarate (Experimental): Patients will switch to tenofovir alafenamide fumarate treatment, 25mg，once a day
  Interventions: Drug: Tenofovir alafenamide fumarate
- Continue with the original regimen (Active Comparator): Patients will continue with the original regimen treatment, entecavir, 0.5mg once a day, or tenofovir disoproxil fumarate 300mg once a day
  Interventions: Drug: Entecavir or Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Tenofovir alafenamide fumarate — Patients would take tenofovir alafenamide fumarate, 25mg，once per day
  Other Names: Vemlidy
  Arms: switch to tenofovir alafenamide fumarate
Drug: Entecavir or Tenofovir disoproxil fumarate — Patients would take entecavir 0.5 mg once per day, or tenofovir disoproxil fumarate 300 mg once per day
  Other Names: Baraclude or Viread
  Arms: Continue with the original regimen

SUMMARY:
Patients with chronic hepatitis B should maximize the inhibition of HBV replication, which could reduce the incidence of liver cancer and liver disease-related complications. However, after 96 weeks of treatment with the first-line drugs, entecavir or tenofovir disoproxil fumarate, a certain proportion of patients still had low levels of HBV replication. Tenofovir alafenamide fumarate is a newly marketed anti-hepatitis B drug that is currently considered to be non-inferior to tenofovir disoproxil fumarate and safer bone and renal effects. Therefore, this research was put forward to investigate whether tenofovir alafenamide fumarate replacement for hepatitis B had a higher virological response rate and safety in patients with low levels of virus after 48 weeks of treatment with entecavir and tenofovir disoproxil fumarate.

DETAILED DESCRIPTION:
Patients who meet the inclusion and exclusion criteria will be enrolled into the research. The participants will voluntarily choose to enter the experimental group or the control group with full informed consent. The control group will continue with the original regimen, while the study group will switch to tenofovir alafenamide fumarate antiviral therapy. Each group will enroll 100 participants.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive for over half a year;
* Age from 18 to 80 years old;
* Entecavir (0.5mg qd) or Tenofovir disoproxil fumarate (300mg qd) for 48 weeks or more;
* HBV DNA level was between 20IU/ ml-2000 IU /mL (COBAS, Taqman).

Exclusion Criteria:

* Low-level viremia of HBV caused by non-standard medication;
* serum total bilirubin is more than 2 times the upper limit of normal (ULN), or ALT or AST is more than 5ULN, or serum albumin is less than 30g/L;
* Overlap with HAV, HCV, HDV, HEV or HIV infection;
* Other liver disease: drug liver disease, alcoholic liver disease, autoimmune liver disease, genetic metabolic liver disease, etc.;
* Decompensated cirrhosis or liver cancer;
* Kidney damage, or autoimmune disease, or other organ failure;
* Combination of Entecavir or Tenofovir disoproxil fumarate ;
* Interferon therapy within half a year;
* Entecavir (0.5mg qd) or Tenofovir disoproxil fumarate;
* Investigator considering inappropriate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Ratio of patients with undetectable hepatitis b virus DNA after treatment | 24 week
  Hepatitis b virus DNA would be tested to know the ratio of patients with undetectable hepatitis b virus DNA at 24 week after treatment.
The changes of glomerular filtration rate | 0 week, 12 week, 24 week, 48 week, 72 week, 96 week, 120 week, 144 week
  Glomerular filtration rate will be tested to know the changes after treatment
The changes of bone mineral density in lumbar spine and hip | 0 week, 48 week, 96 week, 144 week.
  Bone mineral density in lumbar spine and hip were tested after treatment

SECONDARY OUTCOMES:
Ratio of patients with undetectable hepatitis b virus DNA after treatment | 12 week, 48 week, 72 week, 96 week, 120 week, 144 week
  Hepatitis b virus DNA would be tested at 6 time points.
The changes of HBsAg | 0 week, 12 week, 24 week, 48 week, 72 week, 96 week, 120 week, 144 week
  The levels of HBsAg were tested at each time point.
The changes of the degree of liver fibrosis | 0 week, 48 week, 96 week, 144 week.
  Fibroscan would be conducted once every 48 weeks
Differences in symptoms | 0 week, 12 week, 24 week, 48 week, 72 week, 96 week, 120 week, 144 week
  Symptoms would be evaluated at each time point
The changes of HBeAg | 0 week, 12 week, 24 week, 48 week, 72 week, 96 week, 120 week, 144 week
  The levels of HBeAg were tested at each time point.
The changes of alanine aminotransferase | 0 week, 12 week, 24 week, 48 week, 72 week, 96 week, 120 week, 144 week
  The levels of alanine aminotransferase were tested at each time point.
Differences in body weight | 0 week, 12 week, 24 week, 48 week, 72 week, 96 week, 120 week, 144 week
  Body weight would be evaluated at each time point
Differences in proteinuria, albuminuria and urinary β2-microglobulin | 0 week, 12 week, 24 week, 48 week, 72 week, 96 week, 120 week, 144 week
  Proteinuria, albuminuria and urinary β2-microglobulin would be evaluated at each time point
Differences in osmotic pressure | 0 week, 12 week, 24 week, 48 week, 72 week, 96 week, 120 week, 144 week
  The levels of osmotic pressure would be evaluated at each time point
Differences in blood calcium and phosphorus | 0 week, 12 week, 24 week, 48 week, 72 week, 96 week, 120 week, 144 week
  The levels of blood calcium and phosphorus would be evaluated at each time point
Differences in blood lipid | 0 week, 12 week, 24 week, 48 week, 72 week, 96 week, 120 week, 144 week
  The levels of blood lipid would be evaluated at each time point
Differences in serum creatine kinase | 0 week, 12 week, 24 week, 48 week, 72 week, 96 week, 120 week, 144 week
  The levels of creatine kinase would be evaluated at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Yuehua Huang, doctorate, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No